CLINICAL TRIAL: NCT00954486
Title: An Open-Label, Single-Arm Pilot Study of the Efficacy of Erythropoietin Alfa in Improving Peak Oxygen Consumption in Elderly Subjects With Unexplained Anemia
Brief Title: Erythropoietin Alfa in Elderly Subjects With Unexplained Anemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in identifying interested subjects.
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stanley L Schrier, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15270; SPO 36101 (Other: Stanford University); SU-01202009-159 (Other: Stanford University)
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epoetin alfa, 10,000 units/week (Experimental): Epoetin alfa is a recombinant erythropoietin.
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — Epoetin alfa will be administered at 10,000 units/week
  Other Names: Epogen; Procrit

SUMMARY:
The primary objective of this study is to assess the ability of epoetin alfa to raise hemoglobin (Hb) levels in elderly outpatients with unexplained anemia. The secondary objectives of this study are to assess the ability of epoetin alfa to improve physical function; cognitive function; and quality of life, and to assess the safety of epoetin alfa in the study population.

DETAILED DESCRIPTION:
Eligible subjects will be recruited out of the companion study "Anemia in the Elderly" (NCT00640172), after active participation in that study is complete. Subjects will have had a full hematologic evaluation, and unexplained anemia will have been previously defined.

Subjects will provide baseline physical function testing, including exercise testing on a treadmill and testing how far patients can walk in 6 minutes (walk test), as well as quality of life; activity level; and mental functioning.

Study visits will be weekly, and the dose level may be adjusted to achieve the target hemoglobin level within 16 weeks. Once at target, the drug will be taken for a total of 12 additional weeks. The maximum time on the study drug could be 28 weeks, and the minimum time be on the 14 weeks.

The walk tests and questionnaires will be repeated when the target hemoglobin level is reached, and when treatment is completed. The tests about quality of life, activity level, and mental functioning will be repeated at the end of treatment. Follow-up visits will be every 4 weeks for 12 weeks to check for side effects.

ELIGIBILITY:
INCLUSION CRITERIA:

* Aged ≥ 65
* Hb ≤ 11 g/dL
* Outpatient at either the VA Palo Alto Health Care Systems (VAPAHCS) or Stanford Hospital and Clinics (SHC)
* Independently living in the community (ie, not institutionalized or living in a group home)
* Ability to understand and the willingness to sign a written informed consent document
* Performance level ECOG 2 or better
* Diagnosis of unexplained anemia

EXCLUSION CRITERIA:

* Substance abuse or mental health or other problems that would affect compliance with the protocol
* Predicted mortality based on co-morbidities of less than 3 months
* On any erythropoiesis-stimulating agent in the prior 3 months
* Known HIV; hepatitis B; or hepatitis C chronic infection
* Clinically significant and uncontrolled medical condition considered a high risk for participation in an investigational study
* Serum albumin < 3 g/dL
* Use of an investigational medication or participation in an investigational study within 4 weeks prior to enrollment in the trial
* Liver disease as defined as total bilirubin ≥ 2 g/dL or AST/ALT ≥ 2 times the upper limit of normal
* Allergy to recombinant human erythropoietin
* Estimated glomerular filtration rate by Modification of Diet in Renal Disease (MDRD) equation of < 30 mL/min/1.73 m2 or dialysis
* History of proximal deep venous thrombosis or pulmonary embolism within the past 12 months
* Known contraindication to exercise testing

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin (Hb) levels | 14 to 28 weeks
  Measured in mg/dL

SECONDARY OUTCOMES:
Improve physical function | 4 to 30 weeks
  Assessed by questionnaire
Improve cognitive function | 16 to 30 weeks
  Assessed by questionnaire
Improve quality of life | 4 to 30 weeks
  Assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stanley L Schrier, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - VAPAHCS, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California
  - The University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No